CLINICAL TRIAL: NCT05179486
Title: Molecular Epidemiology of Biliary Tree Cancers
Status: Recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-0089
Record Dates: First submitted 2021-12-13; First posted 2022-01-05 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Cholangiocarcinoma; Malignant Digestive System Neoplasm
MeSH Terms: conditions — Cholangiocarcinoma; Gastrointestinal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational (biospecimen collection, questionnaire): Participants complete a questionnaire over 20 minutes. Participants also undergo collection of blood and leftover tissue samples.
  Interventions: Procedure: Biospecimen Collection; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of tissue, and blood
  Other Names: Biological Sample Collection; Biospecimen Collected
Other: Questionnaire Administration — Complete questionnaire

SUMMARY:
This study is to learn if certain risk factors (environmental, viral, behavioral, medical, and dietary), tumor markers, and genetic changes can predict the development and outcome of biliary tree cancers. Establishing biomarkers models from patients may help doctors to further understand how biliary tree cancer is affected by different treatments, and why some people's cancer responds differently than others.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To identify significant factors that may contribute to the etiology of biliary tree cancer.

II. To identify novel genetic loci that predispose to gallbladder cancers (GBC) and cholangiocarcinoma (CGC) diagnosis.

EXPLORATORY AND CORRELATIVE OBJECTIVES:

I. To use the collected blood and tissue materials for exploratory analysis to identify markers that predict prognosis of biliary tree cancers.

II. To correlate the identified markers with results of specific aim I and II to test the interaction between the identified markers with environmental and genetic factors.

OUTLINE:

Participants complete a questionnaire over 20 minutes. Participants also undergo collection of blood and leftover tissue samples.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically or radiologically confirmed diagnosis of CGC or GBC
* With or without prior radiation or chemotherapy
* All United States of America (USA) and non USA residents
* No age, gender, or racial restriction
* Healthy control with no current or history of cancer
* Healthy controls are USA and non USA residents
* Healthy controls are matched to the cases in age (5 years), gender, and race
* Healthy controls are friends and spouses of patients with other than gastro-intestinal (GI) cancers
* Chronic Liver Disease (CLD) controls with no current or history of cancer
* CLD controls are USA and non USA residents
* CLD controls are frequency matched to CGC cases by age (5 years), gender, and race
* CLD controls are patients are diagnosed with or without liver biopsy (core or fine needle aspiration)
* CLD controls must not have evidence liver cancer diagnosis by computed tomography (CT) or magnetic resonance imaging (MRI)

Exclusion Criteria:

* None

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients with biliary tree cancer and healthy participants
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2017-09-25 (Actual); Primary Completion 2027-02-02 (Estimated); Study Completion 2027-02-02 (Estimated)

PRIMARY OUTCOMES:
Significant factors that may contribute to the etiology of biliary tree cancer | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Manal M Hassan, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center website — http://www.mdanderson.org